CLINICAL TRIAL: NCT00405366
Title: A Pilot Neoadjuvant Clinical Trial With Evaluation of Molecular Effects With Sorafenib Tosylate for Patients With Stage II or Greater Renal Cell Carcinoma
Brief Title: Sorafenib in Treating Patients Undergoing Surgery for Stage II, Stage III, or Stage IV Kidney Cancer
Acronym: NRR
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Doris Duke Charitable Foundation (Other); Bayer (Industry); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0603; CDR0000550127 (Other: PDQ number)
Record Dates: First submitted 2006-11-28; First posted 2006-11-30 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Kidney Cancer
Keywords: stage II renal cell cancer; stage III renal cell cancer; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm Study (Other)
  Interventions: Drug: sorafenib tosylate

INTERVENTIONS:
Drug: sorafenib tosylate — Patients will receive treatment with 400mg of sorafenib, orally, twice daily, on a continuous basis as a single agent for at least 4 weeks, but not more than 8 weeks prior to their scheduled nephrectomy

SUMMARY:
RATIONALE: Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving sorafenib before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This clinical trial is studying the side effects and how well sorafenib works in treating patients undergoing surgery for stage II, stage III, or stage IV kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and feasibility of systemic sorafenib tosylate therapy when given prior to definitive nephrectomy in patients with stage II-IV renal cell carcinoma (RCC).

Secondary

* Determine all levels of response in primary renal tumors of patients treated with this drug.
* Assess effects of this drug on gene expression, protein expression, and metabolic profile using tumor tissue samples from these patients.
* Identify biomarkers or biomarker patterns associated with RCC or this drug in these patients.

OUTLINE: This is a pilot, open-label, nonrandomized study.

Patients receive oral sorafenib tosylate twice daily for 4-8 weeks in the absence of disease progression or unacceptable toxicity. After completion of neoadjuvant therapy, patients undergo surgical resection of their kidney tumor.

Patients undergo blood and urine sample collection at baseline and after completion of treatment (i.e., at 4 and 8* weeks) for VEGF analysis. Samples are examined by enzyme-linked immunosorbent assay for measurement of serum and urinary VEGF levels.

NOTE: *Blood sampling at 8 weeks is only for those patients undergoing 8 weeks of study therapy.

Patients also undergo tissue sample collection at the time of nephrectomy. Tissue samples are examined by microarray analysis and IHC staining for expression of CD31/PECAM, HIF1α, and HIF2α. Immunohistochemical staining to identify biomarkers of microvessel density is also performed. Tissue samples are also examined for gene expression and metabolic profile by small molecule mass spectroscopy, as well as VHL gene mutation by VHL mutation analysis.

Patients are followed at 4-8 weeks after nephrectomy.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of renal cell carcinoma (RCC) as confirmed by either of the following:

  * Radiographic documentation by MRI or CT scan
  * Histological evidence of primary RCC
* Stage II-IV disease, as defined by any of the following:

  * T > 7 cm
  * Renal vein involvement
  * Local invasion
  * Evidence of lymph node involvement
  * Distant metastatic disease
* Deemed suitable for nephrectomy by a urologist

  * No requirement for surgery earlier than 4 weeks from study entry
* No known brain metastasis

  * Patients with neurological symptoms must undergo a CT scan or brain MRI to exclude brain metastasis

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Hemoglobin ≥ 9.0 g/dL
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT and AST ≤ 2.5 times ULN (≤ 5 times ULN for patients with liver involvement)
* Creatinine ≤ 2.5 times ULN or glomerular filtration rate ≥ 50 mL/min
* INR ≤ 1.5 AND PTT normal

  * Stable INR required at baseline for patients on warfarin
* Not pregnant or nursing
* Negative pregnancy test
* Fertile women must use effective contraception
* Fertile men must use effective contraception during and for ≥ 2 months after the last dose of sorafenib tosylate
* No other active primary malignancy except skin cancer
* No active coronary artery disease
* No active bleeding diathesis

  * Closely monitored therapeutic anticoagulation allowed
* No cardiac disease, including any of the following:

  * New York Heart Association class III-IV congestive heart failure
  * Unstable angina (i.e., anginal symptoms at rest) or new onset angina (i.e., beginning within the past 3 months)
  * Myocardial infarction within the past 6 months
* No cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* No uncontrolled hypertension, defined as systolic blood pressure (BP) > 150 mm Hg or diastolic BP > 90 mm Hg, despite optimal medical management
* No known HIV infection or chronic hepatitis B or C
* No active, clinically serious infection > grade 2
* No thrombolic or embolic events, such as a cerebrovascular accident or transient ischemic attacks, within the past 6 months
* No pulmonary hemorrhage or bleeding event ≥ grade 2 within the past 4 weeks (≥ grade 3 for any nonpulmonary hemorrhage or bleeding event)
* No serious nonhealing wound, ulcer, or bone fracture
* No significant traumatic injury within the past 4 weeks
* No known or suspected allergy to sorafenib tosylate or any agent given in the course of this study
* No condition that impairs the patient's ability to swallow whole pills
* No malabsorption problem

PRIOR CONCURRENT THERAPY:

* No major surgery or open biopsy within the past 4 weeks
* Concurrent anticoagulation therapy (e.g., warfarin or heparin) allowed
* No other concurrent investigational or commercial agents or therapies for RCC
* No concurrent Hypericum perforatum (St. John's wort) or rifampin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-11; Primary Completion 2009-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Number of subjects experiencing adverse events while taking sorafenib prior to nephrectomy | 8 weeks
  Adverse events will be assessed (graded) using CTCAE criteria
Feasibility of neoadjuvant systemic therapy prior to nephrectomy | 8 weeks
  Feasibility will be measured by the proportion of patients who complete therapy

SECONDARY OUTCOMES:
Response in primary renal tumors | 8 weeks
  All patients will undergo pre and post-treatment tumor imaging by CT or MRI. Measurement of the primary tumor, and up to three largest index lesions for patients with metastatic disease, will be recorded on the case report form. The overall percentage of change in the sum of greatest dimension(s) of the kidney lesion (and three largest index lesions, if any) will be recorded. Response to therapy will be measured in absolute size change, as well as according to traditional RECIST criteria.
Effects of sorafenib tosylate therapy on gene expression, protein expression, and metabolic profile | 8 weeks
  Microarray data will be done using statistical analysis and hierarchical clustering with the assistance of the UNC Genomics and Bioinformatics Core Facility

CONTACTS AND LOCATIONS:
Overall Officials: W. Kimryn Rathmell, MD, PhD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States